CLINICAL TRIAL: NCT02544776
Title: Effect of Amlodipine and Clomid on Blood Flow of Preovulatory Follicle in Polycystic Ovarian Patients
Brief Title: Amlodipine on Blood Flow of Preovulatory Follicle in Polycystic Ovarian Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Fathy Ali Mohamed Ghanem (Other)
Responsible Party: Sponsor-Investigator, Ahmed Fathy Ali Mohamed Ghanem, Resident of Obstetrics and Gynecology, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: effect of amlodipine in pco
Record Dates: First submitted 2015-08-27; First posted 2015-09-09 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Female Infertility Associated With Anovulation
Keywords: pco; Amlodipine
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Clomiphene; Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clomifene citrate and Amlodipine (Experimental): Amlodipine 5mg tablet and Clomifene citrate 50 mg tablet once by mouth daily at morning starting from day number 5 of menstrual cycle till day number 9.
  Interventions: Drug: Clomifene citrate ( clomid 50 mg ); Drug: Amlodipine
- Clomifene citrate (Active Comparator): Clomifene citrate 50mg and once daily at morning starting from day number 5 of menstrual cycle till day number 9
  Interventions: Drug: Clomifene citrate ( clomid 50 mg )

INTERVENTIONS:
Drug: Clomifene citrate ( clomid 50 mg )
  Other Names: clomid ( 50 mg )
Drug: Amlodipine
  Other Names: Norvasc 5mg
  Arms: Clomifene citrate and Amlodipine

SUMMARY:
On the basis of the current study, amlodipine seems to be a promising drug on improving uterine, ovarian blood flow, size of pre-ovulatory follicle, midluteal progesterone level and pregnancy outcome in patients with pco.

DETAILED DESCRIPTION:
To know if amlodipine has vasodilator effect on ovarian ar. In pco patient.

ELIGIBILITY:
Inclusion Criteria:

* Demographic features including females in age of ≥20 & ≤35, and BMI of ≤39.
* Infertility secondary to polycystic ovary , The choice of polycystic ovary patients will be according to the Rotterdam consensus workshop (Rotterdam, 2004), and the diagnosis of polycystic ovary by ultrasonography will be made according to Adams et al. criteria which are the most often cited (Adams et al., 1985).The Rotterdam criteria as follows:

  * Oligo- or anovulation.
  * Clinical and/or biochemical signs of hyper androgynism
  * The presence of polycystic ovaries on ultrasound scan. Ultrasound findings of enlarged ovaries with multiple small cysts (10-12 or more of 2-9 mm in diameter) scattered around the periphery and highly echogenic stroma

Exclusion Criteria:

* Including other causes of infertility diagnosed during infertility work up.
* Patients refused to participate or to continue study.
* Also, hepatic, cardiac, and hypotensive patients will be excluded from the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
change in ovarian artery perfusion | day number five and day number 9 of menstrual cycle
  peak systolic velocity ( psv ) measured by doppler u/s

SECONDARY OUTCOMES:
Number of mature follicle | day 14 of menstrual cycle
  by vaginal u/s
endometrial thickening | day number five and day number 9 of menstrual cycle
  by vaginal u/s